CLINICAL TRIAL: NCT00569478
Title: The Effect of Rehabilitation for Patients Living With an ICD
Brief Title: The Effect of Rehabilitation for Patients Living With an Implantable Cardioverter Defibrillator
Acronym: ICD-rehab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Selina Kikkenborg Berg, Ph.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-Berg
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Quality of Life
Keywords: ICD; Rehabilitation
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): rehabilitation
  Interventions: Other: rehabilitation
- 2 (No Intervention): controls

INTERVENTIONS:
Other: rehabilitation — Nursing consultations and physical training
  Arms: 1

SUMMARY:
The purpose of this study is to describe the effect and meaning of an outpatient-nursing programme including physical activity for patients with implantable cardioverter defibrillators (ICD).

Hypothesis: The outpatient nursing programme will increase the perceived health and quality of life; improve the management of life from a patient perspective; reduce fear of exercise and increase physical capability and reduce the number of treatment-demanding arrhythmias.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillators (ICD) are used in the treatment of life-threatening heart arrhythmia and the prevention of sudden cardiac death (SCD). The ICD terminates arrhythmia by delivering therapy in the form of electrical impulses to the heart. Patients have described the high energy shock administered by the devise as feeling like a painful kick in the chest.

Patients, who receive an ICD are very much protected against SCD and it is assumed that they are less worried and effected by their heart disease than others. That is not correct though. Studies have shown, that living with an ICD can lead to anxiety, fear of shock and avoidance of situations, places and objects that are associated to shock. It often leads to social isolation, avoidance of physical activity and mood-disturbances.

The purpose of this study is to describe the effect and meaning of an outpatient-nursing programme including physical activity for patients with ICD.

Hypothesis: see above

Intervention: The outpatient nursing programme has a duration of 1 year and is directed towards parameters that ICD reportedly affect. The focus is prevention of the known risks and problems. The content is partly information and education in managing an ICD, partly emotional reactions and further discussion of handling life with ICD. 3-month into the program physical training lead by a physical therapist is started. It is optimal whether to carry out the twice-weekly physical training program at home or at the hospital.

180 patients, who get an ICD transplanted at Copenhagen university Hospital, Rigshospitalet, are included in the study prior to discharge. 90 patients in the intervention group and 90 controls.

Using questionnaires, qualitative interviews, work-test, 6 MWT and decoding ICD the effect and meaning of the programme is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* In-patients at Copenhagen University Hospital who just received an ICD for the first time.

Exclusion Criteria:

* Patients who:

  * do not understand the instructions,
  * are under 18 years old,
  * are diagnosed with a mental disease,
  * suffer from a competing disease,
  * can not participate in physical training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | 3 -6-12 month
Physical capability | 3-6-12 month

CONTACTS AND LOCATIONS:
Overall Officials: Selina K Berg, PhD Fellow, Principal Investigator — Rigshospitalet, Denmark; Jesper H Svendsen, Principal Investigator — Rigshospitalet, Denmark; Preben U Pedersen, Principal Investigator — Aarhus Universitet; Birthe D Pedersen, Principal Investigator — Aarhus Universitet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Berg SK, Moons P, Zwisler AD, Winkel P, Pedersen BD, Pedersen PU, Svendsen JH. Phantom shocks in patients with implantable cardioverter defibrillator: results from a randomized rehabilitation trial (COPE-ICD). Europace. 2013 Oct;15(10):1463-7. doi: 10.1093/europace/eut087. Epub 2013 Apr 18. PMID 23599170
- [Derived] Berg SK, Svendsen JH, Zwisler AD, Pedersen BD, Preisler P, Siersbaek-Hansen L, Hansen MB, Nielsen RH, Pedersen PU. COPE-ICD: a randomised clinical trial studying the effects and meaning of a comprehensive rehabilitation programme for ICD recipients -design, intervention and population. BMC Cardiovasc Disord. 2011 Jun 17;11:33. doi: 10.1186/1471-2261-11-33. PMID 21682864